CLINICAL TRIAL: NCT04858464
Title: Reliability, Validity, and Cross-Cultural Adaptation of the Turkish Version of the Primary Sjögren Syndrome Quality of Life (PSS-QoL) Questionnaire
Brief Title: Reliability, Validity of the Turkish Version of the Primary Sjögren Syndrome Quality of Life (PSS-QoL) Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selin Bayram, Msc, Gazi University
Other Study IDs: E-77082166-604.01.02-27503
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's Syndrome; Quality of Life; Patient-reported Outcome; Reliability; Validity
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Individuals with primary Sjögren's syndrome
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Patients will complete the mentioned questionnaires.
  Other Names: Questionnaire application

SUMMARY:
The purpose of this study was to investigate adaptation, validity, and reliability of the Turkish version of the Primary Sjögren's Syndrome Quality of Life (PSS-QoL) Questionnaire

DETAILED DESCRIPTION:
Primary Sjögren's Syndrome (PSS) is a chronic systemic disease characterized by lymphocytic infiltration of exocrine glands. Dryness, chronic pain, physical fatigue, glandular and extraglandular symptoms seen in PSS cause deterioration of the health-related quality of life.

The Primary Sjögren's Syndrome Quality of Life (PSS-QoL) Questionnaire has recently developed as a patient-reported condition-specific outcome measurement tool to assess the quality of life associated with PSS. The PSS-QoL questionnaire consists of 25 questions with a physical and psychosocial dimension.The physical dimension consists of a numeric rating scale (NRS, ranging from 0 to 10) for pain and physical symptoms. The question related to vaginal dryness is intended to be answered by women only. Each "yes" answer about physical symptoms-related questions adds 1 point to the score. The psychosocial dimension can be scored on a 5-point Likert scale and contains 14 question with the following possible answers: never (0), rarely (1), sometimes (2), often (3), and always (4). The PSS-QoL score ranges from 0-96 (for women) and 0-92 (excluding the question of vaginal dryness for men). After questioning the sociodemographic characteristics of the individuals, PSS-QoL, EuroQuol-5D, the EULAR Sjögren's Syndrome Disease Activity Index and EULAR Sjögren's Syndrome Patient Reported Index will be used. Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary Sjögren's syndrome

Exclusion Criteria:

* Having neurological and cognitive disorders,
* Having another rheumatological diseases

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary Sjögren's syndrome between the ages of 18-90
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-05-02 (Estimated)

PRIMARY OUTCOMES:
Primary Sjögren's Syndrome Quality of Life (PSS-QoL) Questionnaire | 10 minutes
  Primary Sjögren's Syndrome Quality of Life (PSS-QoL) Questionnaire was designed to evaluate measurement of health related quality of life in patients with primary Sjögren's syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Assoc. Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lackner A, Stradner MH, Hermann J, Unger J, Stamm T, Graninger WB, Dejaco C. Assessing health-related quality of life in primary Sjogren's syndrome-The PSS-QoL. Semin Arthritis Rheum. 2018 Aug;48(1):105-110. doi: 10.1016/j.semarthrit.2017.11.007. Epub 2017 Nov 27. PMID 29395257
- [Background] Ng WF, Bowman SJ. Primary Sjogren's syndrome: too dry and too tired. Rheumatology (Oxford). 2010 May;49(5):844-53. doi: 10.1093/rheumatology/keq009. Epub 2010 Feb 10. PMID 20147445
- [Background] Lackner A, Ficjan A, Stradner MH, Hermann J, Unger J, Stamm T, Stummvoll G, Dur M, Graninger WB, Dejaco C. It's more than dryness and fatigue: The patient perspective on health-related quality of life in Primary Sjogren's Syndrome - A qualitative study. PLoS One. 2017 Feb 9;12(2):e0172056. doi: 10.1371/journal.pone.0172056. eCollection 2017. PMID 28182787